CLINICAL TRIAL: NCT03252535
Title: Dose-Response Evaluation of the Investigational Product Cellavita HD After Intravenous Administration in Patients With Huntington's Disease
Brief Title: Dose-response Evaluation of the Cellavita HD Product in Patients With Huntington's Disease
Acronym: ADORE-DH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Cellavita Pesquisa Científica Ltda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADORE-DH; 52375916.1.0000.5412 (Other: CAAE)
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Huntington Disease
Keywords: Huntington disease; Stem cell therapy; Dental pulp stem cell
MeSH Terms: conditions — Huntington Disease | interventions — Cell- and Tissue-Based Therapy; Cell Count

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study drugs will be provided in identical packages to maintain the study masking. Neither the Investigator nor the study team will know which drug the subject is receiving. In addition, the external outcome evaluator will receive the results in a codified manner (concealed).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cellavita HD Lower Dose (Experimental): The participants randomized to this group will receive a total of 9 intravenous administrations of 1x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 120 days (total of 3 cycles).
  Interventions: Biological: Cellavita HD lower dose
- Cellavita HD Higher Dose (Experimental): The participants randomized to this group will receive a total of 9 intravenous administrations of 2x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 120 days (total of 3 cycles).
  Interventions: Biological: Cellavita HD higher dose
- Placebo Group (Placebo Comparator): The participants randomized to this group will receive a total of 9 intravenous administrations divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 120 days (total of 3 cycles).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Cellavita HD lower dose — The participants will receive a total of 9 intravenous administrations of 1x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 120 days (total of 3 cycles).
  Other Names: cellular therapy, mesenchymal stem cells
  Arms: Cellavita HD Lower Dose
Biological: Cellavita HD higher dose — The participants will receive a total of 9 intravenous administrations of 2x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 120 days (total of 3 cycles).
  Other Names: cellular therapy, mesenchymal stem cells
  Arms: Cellavita HD Higher Dose
Other: Placebo — The participants will receive a total of 9 intravenous administrations of placebo divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 120 days (total of 3 cycles).
  Other Names: physiological solution without cells
  Arms: Placebo Group

SUMMARY:
Cellavita HD is a stem-cell therapy for Huntington's Disease. This is a prospective, phase II, single-center, randomized (2:2:1), triple-blind, placebo controlled study, with two test doses of Cellavita HD product.

DETAILED DESCRIPTION:
This is a phase II dose-response study in which participants with HD will receive three intravenous injections of the investigational product or placebo (one every month for three months) a total of three cycles. The subjects will be randomized in 2: 2: 1 ratio for the groups G1: lower dose (1x10^6 cells/weight range), G2: higher dose (2x10^6 cells/weight range) or G3: placebo. To identify the dose of the product that will provide the best clinical response, motor assessment will be performed with UHDRS scale and improvement will be evaluated by correlating before and after treatment scores. Additionally, also will be performed the combined score through the cUHDRS. Secondary evidences of efficacy will be evaluated through the data of functional state, total functional capacity, functional independence, psychiatric symptoms and cognition from UHDRS scale. Additionally, related data to clinical worsening, change of Body Mass Index (BMI), risk of suicide attempt and neurological image improvement will be evaluated. Safety evaluation will included the incidence and classification of the adverse events experienced by the subjects during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide a written, signed and dated Informed Consent Form;
2. Male and female subjects aged ≥ 21 and ≤ 65 years;
3. Have a confirmatory diagnosis report (PCR) of Huntington's disease with a number of CAG repeats in chromosome 4 higher than or equal to 40, and lower than or equal to 50 (if the subject did not perform the exam and/or if he/she does not have an available result for this exam, a new exam must be performed);
4. A score of 5 points or higher for the motor evaluation of the UHDRS scale (Unified Huntington's Disease Rating Scale) at enrollment;
5. Score of 8 to 11 points for the functional capacity of the UHDRS scale at enrollment.

Exclusion Criteria:

1. Subject who participated in clinical trials protocols within the last twelve (12) months (Resolution CNS 251, August 7, 1997, item III, subitem J), unless, at the investigator's opinion, the subject would have a direct benefit from it;
2. Diagnosis of juvenile Huntington's disease;
3. Diagnosis of epilepsy;
4. Diagnosis of major cognitive disorder;
5. Active decompensated psychiatric illness;
6. Current or prior history of neoplasm;
7. Current history of gastrointestinal, hepatic, renal, endocrine, pulmonary, hematological, immunological, metabolic pathology or severe uncontrolled cardiovascular diseases;
8. Diagnosis of any active infection, whether viral, bacterial, fungal or caused by another pathogen;
9. Subject with contraindication to the exams performed in this study, for example, with pacemaker or surgical clip; Alcohol and drugs abuse (previously diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders - DSM V criteria);
10. Use of illegal drugs;
11. Tabagism;
12. Smoker or quit smoking for less than 6 months;
13. Positive result in one of the serum tests: HIV 1 and 2 (Anti-HIV-1,2), HTLV I and II, HBV (HBsAg, Anti-HBc), HCV (anti-HCV-Ab) and FTA-ABS (Treponema pallidum);
14. History of drug allergy, including to contrast agents used in imaging tests or bovine-derived products;
15. Using or expects to use immunosuppressant drugs or forbidden drugs (item 5.3) during the first three months after the first administration of the investigational product;
16. Any clinical change that the investigator considers a risk to subject's enrollment in the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Macedo da Silva, MD, Principal Investigator — Azidus Brasil Scientific Research and Development Ltda
Locations (1):
- Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data will become public.

REFERENCES:
- [Background] Aleynik A, Gernavage KM, Mourad YSh, Sherman LS, Liu K, Gubenko YA, Rameshwar P. Stem cell delivery of therapies for brain disorders. Clin Transl Med. 2014 Jul 19;3:24. doi: 10.1186/2001-1326-3-24. eCollection 2014. PMID 25097727
- [Background] de Almeida FM, Marques SA, Ramalho Bdos S, Rodrigues RF, Cadilhe DV, Furtado D, Kerkis I, Pereira LV, Rehen SK, Martinez AM. Human dental pulp cells: a new source of cell therapy in a mouse model of compressive spinal cord injury. J Neurotrauma. 2011 Sep;28(9):1939-49. doi: 10.1089/neu.2010.1317. Epub 2011 Aug 8. PMID 21609310
- [Background] Barker RA, Mason SL, Harrower TP, Swain RA, Ho AK, Sahakian BJ, Mathur R, Elneil S, Thornton S, Hurrelbrink C, Armstrong RJ, Tyers P, Smith E, Carpenter A, Piccini P, Tai YF, Brooks DJ, Pavese N, Watts C, Pickard JD, Rosser AE, Dunnett SB; NEST-UK collaboration. The long-term safety and efficacy of bilateral transplantation of human fetal striatal tissue in patients with mild to moderate Huntington's disease. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):657-65. doi: 10.1136/jnnp-2012-302441. Epub 2013 Jan 23. PMID 23345280
- [Background] Bonelli RM, Wenning GK. Pharmacological management of Huntington's disease: an evidence-based review. Curr Pharm Des. 2006;12(21):2701-20. doi: 10.2174/138161206777698693. PMID 16842168
- [Background] de Souza PV, Alves FB, Costa Ayub CL, de Miranda Soares MA, Gomes JR. Human immature dental pulp stem cells (hIDPSCs), their application to cell therapy and bioengineering: an analysis by systematic revision of the last decade of literature. Anat Rec (Hoboken). 2013 Dec;296(12):1923-8. doi: 10.1002/ar.22808. Epub 2013 Oct 15. PMID 24130093
- [Background] Fink KD, Deng P, Torrest A, Stewart H, Pollock K, Gruenloh W, Annett G, Tempkin T, Wheelock V, Nolta JA. Developing stem cell therapies for juvenile and adult-onset Huntington's disease. Regen Med. 2015;10(5):623-46. doi: 10.2217/rme.15.25. PMID 26237705
- [Background] Kerkis I, Caplan AI. Stem cells in dental pulp of deciduous teeth. Tissue Eng Part B Rev. 2012 Apr;18(2):129-38. doi: 10.1089/ten.TEB.2011.0327. Epub 2011 Dec 28. PMID 22032258
- [Background] Ross CA, Aylward EH, Wild EJ, Langbehn DR, Long JD, Warner JH, Scahill RI, Leavitt BR, Stout JC, Paulsen JS, Reilmann R, Unschuld PG, Wexler A, Margolis RL, Tabrizi SJ. Huntington disease: natural history, biomarkers and prospects for therapeutics. Nat Rev Neurol. 2014 Apr;10(4):204-16. doi: 10.1038/nrneurol.2014.24. Epub 2014 Mar 11. PMID 24614516
- [Background] Kaplan A, Stockwell BR. Therapeutic approaches to preventing cell death in Huntington disease. Prog Neurobiol. 2012 Dec;99(3):262-80. doi: 10.1016/j.pneurobio.2012.08.004. Epub 2012 Aug 28. PMID 22967354
- [Background] Weiss A, Trager U, Wild EJ, Grueninger S, Farmer R, Landles C, Scahill RI, Lahiri N, Haider S, Macdonald D, Frost C, Bates GP, Bilbe G, Kuhn R, Andre R, Tabrizi SJ. Mutant huntingtin fragmentation in immune cells tracks Huntington's disease progression. J Clin Invest. 2012 Oct;122(10):3731-6. doi: 10.1172/JCI64565. Epub 2012 Sep 17. PMID 22996692
- [Background] Langbehn DR, Brinkman RR, Falush D, Paulsen JS, Hayden MR; International Huntington's Disease Collaborative Group. A new model for prediction of the age of onset and penetrance for Huntington's disease based on CAG length. Clin Genet. 2004 Apr;65(4):267-77. doi: 10.1111/j.1399-0004.2004.00241.x. PMID 15025718
- [Derived] Fernandes JMS, Pagani E, Wenceslau CV, Ynoue LH, Ferrara L, Kerkis I. Phase II trial of intravenous human dental pulp stem cell therapy for Huntington's disease: a randomized, double-blind, placebo-controlled study. Stem Cell Res Ther. 2025 Aug 6;16(1):432. doi: 10.1186/s13287-025-04557-2. PMID 40770775
- [Derived] Wenceslau CV, de Souza DM, Mambelli-Lisboa NC, Ynoue LH, Araldi RP, da Silva JM, Pagani E, Haddad MS, Kerkis I. Restoration of BDNF, DARPP32, and D2R Expression Following Intravenous Infusion of Human Immature Dental Pulp Stem Cells in Huntington's Disease 3-NP Rat Model. Cells. 2022 May 17;11(10):1664. doi: 10.3390/cells11101664. PMID 35626701

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 49 enrolled participants, 35 met the inclusion criteria and were randomized to treatment.
Groups:
- Nestacell (Former Cellavita HD) Lower Dose: The participants randomized to this group will receive a total of 9 intravenous administrations of 1x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycle every 120 days (a total of 3 cycles).
  NestaCell lower dose: The participants will receive a total of 9 intravenous administrations of 1x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycle every 120 days (a total of 3 cycles).
- Nestacell (Former Cellavita HD) Higher Dose: The participants randomized to this group will receive a total of 9 intravenous administrations of 2 × 10^6 cells/weight range, divided into three administrations per cycle. Each administration will occur every 30 days and cycle every 120 days (a total of 3 cycles).
  NestaCell higher dose: The participants will receive a total of 9 intravenous administrations of 2x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycle every 120 days (a total of 3 cycles).
Period: Overall Study
Arm/Group | Nestacell (Former Cellavita HD) Lower Dose | Nestacell (Former Cellavita HD) Higher Dose | Placebo Group
Started | 14 | 14 | 7
Completed | 13 | 12 | 7
Not Completed | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Met discontinuation criteria | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nestacell (Former Cellavita HD) Lower Dose | Nestacell (Former Cellavita HD) Higher Dose | Placebo Group | Total
Number analyzed (Participants) | 14 | 14 | 7 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (9.4) | 43.7 (8.5) | 50.9 (9.7) | 48.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 2 | 18
  Male | 7 | 5 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 2 | 1 | 0 | 3
  Multiracial | 3 | 3 | 3 | 9
  White | 9 | 9 | 4 | 22
  Other | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 14 | 14 | 7 | 35
Height [Mean (Standard Deviation); unit: meters] | 1.63 (0.08) | 1.61 (0.1) | 1.66 (0.06) | 1.63 (0.08)
Weight [Mean (Standard Deviation); unit: Kg] | 65.5 (14.0) | 68.7 (14.5) | 69.3 (14.0) | 67.8 (14.2)
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 24.4 (4.5) | 26.4 (5.5) | 25.0 (4.4) | 25.3 (4.8)
CAG repeat [Count of Participants; unit: Participants]
  <44 | 9 | 7 | 4 | 20
  >=44 | 5 | 7 | 3 | 15
CAP scale [Mean (Standard Deviation); unit: units on a scale] — The CAP scale (CAG-Age Product) measures cumulative disease burden in Huntington's disease by multiplying age by the difference between CAG repeat length and 35.5. Scores range from 0 to over 100, with higher values indicating greater genetic exposure, higher risk, and closer proximity to symptom onset (CAP=100 approximates average motor diagnosis age). It is a single composite score (units on a scale); lower scores indicate better outcomes, higher scores worse.
  units on a scale | 106.7 (18.6) | 97.5 (11.5) | 110.7 (12.0) | 105.0 (14.0)
Years of symptoms [Mean (Standard Deviation); unit: years] | 10.1 (3.6) | 7.4 (2.1) | 10.1 (3.2) | 9.2 (3.0)
UHDRS Total Motor Score [Mean (Standard Deviation); unit: units on a scale] — The Unified Huntington's Disease Rating Scale Total Motor Score (UHDRS-TMS) is a clinician-rated scale assessing motor symptoms in Huntington's disease. It comprises 31 items grouped in 15 domains, such as chorea, dystonia, rigidity, oculomotor function, balance, and others. Scores range from 0 (normal motor function) to 124 (worst impairment). Higher scores indicate worse motor function and more severe disease progression. The total motor score is computed by summing the item scores on a 0-4 severity scale, resulting in a composite summed score measured in units on a scale.
  units on a scale | 43.6 (23.8) | 20.7 (11.8) | 38.0 (7.5) | 34.1 (14.4)
UHDRS Total Functional Capacity [Mean (Standard Deviation); unit: units on a scale] — The Unified Huntington's Disease Rating Scale Total Functional Capacity (UHDRS-TFC) assesses a person's ability to manage work, finances, daily living, domestic chores, and care needs in Huntington's disease. It is a sum score of 5 items, with a range from 0 to 13, where higher scores indicate better functional capacity and lower scores reflect worse functioning or greater disability. The total score is computed by summing points from each item, measured in units on a scale.
  units on a scale | 8.1 (2.1) | 8.4 (2.6) | 6.7 (1.4) | 7.7 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy by UHDRS-TMS
Description: The primary endpoint was the rate of change (slope) in Unified Huntington's Disease Rating Scale - Total Motor Score from V0 to V11 (minimum 0, the best; and maximum 124, the worst). For each participant, a regression line was fitted (Y = a + bx), where b represents the individual slope, reflecting the annualised rate of motor progression. A negative slope suggests improvement or slower decline; a positive slope indicates worsening. To compare treatment efficacy, the slopes were analysed using a Mixed Model for Repeated Measures (MMRM), which accounts for intra-subject variability and missing data. This approach allowed estimation and comparison of average slopes between each treated group and placebo, providing a robust measure of motor function trajectory over time.
Time Frame: monthly for eleven months
Measure: Mean (Standard Error); unit: score on a scale/year
Arm/Group | Nestacell (Former Cellavita HD) Lower Dose | Nestacell (Former Cellavita HD) Higher Dose | Placebo Group
Number analyzed (Participants) | 14 | 14 | 7
score on a scale/year | -1.23 (0.84) | 0.84 (0.90) | 8.91 (1.11)

2. Secondary Outcome: Efficacy by UHDRS-TFC
Description: Assessed by the rate of change (slope) from V0 to V11 in the UHDRS-TFC.
  The response of each participant or means of all participants was evaluated by the slopes of each regression line of UHDRS-TFC determined as follows:
  The equation describes the regression line: Y = a + bx, where:
  * "Y" is the dependent variable.
  * "a" is the constant that represents the intersection of the line with the vertical axis.
  * "b" is the angular coefficient, that is, the slope.
  * "x" is the independent variable. Therefore, the 'b' value represents the slope of the straight line that best fits the values collected from the baseline (V0) to the value of V11, using the least squares method. This slope corresponds to the estimated annualized individual variation of UHDRS-TFC during the given period.
Time Frame: monthly for eleven months
Measure: Mean (Standard Error); unit: score on a scale/year
Arm/Group | Nestacell (Former Cellavita HD) Lower Dose | Nestacell (Former Cellavita HD) Higher Dose | Placebo Group
Number analyzed (Participants) | 14 | 14 | 7
score on a scale/year | -0.29 (0.18) | 0.73 (0.18) | -0.89 (0.26)

3. Other Pre Specified Outcome: Exposure to NestaCell (Former Cellavita HD) Product
Description: Number of administrations of NestaCell (Former Cellavita HD) and Placebo
Time Frame: eleven months
Measure: Mean (Standard Deviation); unit: number os adminstrations
Arm/Group | Nestacell (Former Cellavita HD) Lower Dose | Nestacell (Former Cellavita HD) Higher Dose | Placebo Group
Number analyzed (Participants) | 14 | 14 | 7
number os adminstrations | 9.0 (0.0) | 8.4 (1.5) | 9.0 (0.0)

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Nestacell (Former Cellavita HD) Lower Dose | Nestacell (Former Cellavita HD) Higher Dose | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 12/14 | 12/14 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nestacell (Former Cellavita HD) Lower Dose (N=14) | Nestacell (Former Cellavita HD) Higher Dose (N=14) | Placebo Group (N=7)
hospitalized for sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nestacell (Former Cellavita HD) Lower Dose (N=14) | Nestacell (Former Cellavita HD) Higher Dose (N=14) | Placebo Group (N=7)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (3) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal hair growth (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Wound (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Subcutaneous hemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Change in hair color (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Atopic dermatitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (2)
Dyslipidemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cervicogenic gourd pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Normochromic and normocytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (3) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis at the administration site (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Compulsion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Altered mood (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Viral conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dengue Fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Increased blood creatinine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
Positive salmonella test (Investigations) | 0 (0) | 0 (0) | 1 (1)
Abnormal temperature perception test (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (7) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Tooth implant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03252535/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT03252535/SAP_001.pdf